CLINICAL TRIAL: NCT00834951
Title: A Prospective Multicenter Phase II Study of MabThera (Rituximab) Plus 2 Weekly CHOP Followed by Low Dose Total Body Irradiation in Elderly Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Adjuvant Low Dose Total Body Irradiation in Elderly Patients With Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Francesco d'Amore/Consultant, Haematology Department, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTBI-NHL-01
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: Diffuse large B-cell lymphoma; Elderly patients; Low dose total body irradiation; RCHOP14
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Low dose total body irradiation — Low dose total body irradiation is given 3 weeks after the end of chemo-immunetherapy in the form of 4 daily fractions 0.2 Gy per fraction to be repeated after 2 weeks of rest

SUMMARY:
The purpose of this study is to determine whether the application of low dose total body irradiation following chemo-immuntherapy in elderly patients with aggressive with non-Hodgkin's lymphoma would be safe and potentially benecicial adjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* previously untreated, pathology verified aggressive non-Hodgkin lymphoma of the diffuse large B-cell type according to the WHO classification. Age between 60 years and 80 years.Positive for an anti-CD20 antibody. Good performance status and normal initial normal blood count.

Exclusion Criteria:

* Patients with previous lymphoma associated with immune suppression of any sort. Diagnosis or history of indolent lymphoma or other malignancies. Marked impairment of any vital organ such as the heart, lung, liver or kidneys.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)